CLINICAL TRIAL: NCT06316362
Title: Efficacy of SMOF Lipid in the Management of Acute Poisoning With Carbamazepine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMOF in carbamazepine toxicity
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-03

CONDITIONS: Acute Poisoning
Keywords: Carbamazepine poisoning; SMOF lipid; lipophilic agents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): The first group constitutes the control group that was administered the standard treatment protocol for carbamazepine toxicity.
  Interventions: Other: Standard treatment for carbamazepine toxicity
- SMOF lipid treated group (Active Comparator): The second group received the SMOF lipid infusion in addition to the standard protocol.
  Interventions: Drug: SMOF lipid 20%

INTERVENTIONS:
Drug: SMOF lipid 20% — SMOF 20%; a blend of (soybean oil, medium chain triglycerides, olive and fish oil) is a new lipid emulsion product that was provided as a bolus dose of 1.5ml/kg for one hour, followed by a maintenance dose of 6 ml/kg for a period of four hours to the active comparator group
  Arms: SMOF lipid treated group
Other: Standard treatment for carbamazepine toxicity — Hypotension was initially treated with isotonic crystalloid; vasopressors were utilised if intravenous fluids failed to restore the hypotension. This was in the form of norepinephrine with a dose of 0.05 μg/kg/min and titrated till reaching the goal mean arterial pressure (>65 mmHg).
  Those experiencing seizures due to CBZ overdose were treated with benzodiazepines (diazepam) at a dose of 10-20 mg. Benzodiazepines are considered allosteric modulators of the gamma-aminobutyric acid channel.
  MDAC (50 grammes every six hours) was given to all patients in the current study. Those with severe poisoning were given the MDAC after securing the airway with a cuffed endotracheal tube
  Arms: control group

SUMMARY:
The goal of the current study was to evaluate whether SMOF lipid administration could be used as an adjuvant therapy to treat acute, moderate-to-severe carbamazepine poisoning.

DETAILED DESCRIPTION:
Among anticonvulsants, carbamazepine (CBZ) is considered one of the most commonly reported poisonings. Carbamazepine (CBZ) was approved for use as a primary anticonvulsant agent following its initial use for trigeminal neuralgia. Further indications for the drug included treatment for bipolar disorder, resistant schizophrenia, and pain syndromes.

The wide availability of carbamazepine increases the potential for overdose, either accidentally or intentionally. The American Association of Poison Control Centres reported 2,562 hazardous exposures to CBZ in 2020. In addition, CBZ was the most commonly used anti-epileptic drug, according to a recent study by the National Centre for Environmental and Clinical Toxicology Research, Cairo, Egypt.

CBZ works by blocking presynaptic voltage-gated sodium channels, thereby inhibiting the release of synaptic glutamate and other neurotransmitters.

Overdose of CBZ is clinically manifested by nystagmus, nausea, dysarthria, ataxia, sedation, delirium, mydriasis, ophthalmoplegia, and myoclonus. The serious clinical problems resulting from large overdoses of CBZ are cardiotoxicity, respiratory depression, apnea, seizures, and coma. Mortality from CBZ poisoning is uncommon.

Because there is no definitive antidote for carbamazepine poisoning, poison control centres recommend supportive therapy based on the patient's clinical condition and multiple-dose activated charcoal (MDAC) as a specific intervention for enhanced elimination. Nevertheless, the elimination of the drug from the body can be prolonged.

The scarcity of physiological antidotes for acute poisonings encourages toxicologists to supplement standard supportive treatment protocols with promising agents that tend to improve morbidity and mortality.

In this context, intravenous lipid emulsions (ILE) are mainly used as a source of energy and essential fatty acids in patients requiring parenteral nutrition. Apart from their nutritional value, lipid emulsion therapy is becoming increasingly popular in critical care settings as a treatment for toxicity with lipophilic agents, particularly when the standard remedies are ineffective.

Following the encouraging outcomes of using ILEs for the treatment of local anaesthetic systemic toxicity, subsequent studies reported the therapeutic effect of ILEs in acute poisonings with other xenobiotics. However, the evidence for the potential effectiveness of ILE in clinical toxicology consists mainly of case reports and experimental studies. In cases of CBZ poisoning, ILE was not evaluated using a randomised control trial (RCT).

ILE may be suitable for the treatment of CBZ toxicity due to its lipid solubility. To the best of our knowledge, the effect of ILE therapy on acute carbamazepine poisoning has not been studied sufficiently.

SMOF 20%, a blend of soybean oil, medium-chain triglycerides, olive oil, and fish oil, is a new lipid emulsion product that has shown better therapeutic results regarding parentral nutrition when compared with traditional ones such as Intralipid® 20%. It has been associated with decreased oxidative injury, improved liver function, and increased antioxidant activity

ELIGIBILITY:
Inclusion Criteria:

The patients were enrolled in the study in accordance with the following:

1. Gender and age: adult symptomatic males and females.
2. Patients were admitted within 12 hours of exposure to the poison.
3. Patients received no prior treatment before admission.
4. Patients with moderate-to-severe carbamazepine poisoning according to the Poisoning Severity Score (PSS)
5. Patients classified as high-risk (HR) with anti-depressant overdose risk assessment (ADORA) criteria.

Exclusion Criteria:

Patients will be excluded if they have any of the following conditions:

1. pregnant and lactating women.
2. Patients with major medical conditions (e.g. diabetes mellitus), cardiovascular disease, renal, or hepatic failure).
3. Patients suffering from hyperlipidemia.
4. Malignancy.
5. Co-ingestion.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Improvement in Conscious Levels Measured by Glasgow Coma Scale (GCS) | participants were monitored within 24 hours from admission to the hospital
  This study evaluates the efficacy of SMOF lipid 20% in improving conscious levels among participants with acute carbamazepine poisoning within 24 hours. Conscious level improvement is assessed using the Glasgow Coma Scale (GCS), a widely recognised tool for neurological assessment. The GCS measures eye opening, verbal response, and motor response, with higher scores indicating better conscious levels. The study aims to determine the extent of improvement in GCS scores following SMOF lipid administration, providing valuable insights into its effectiveness in enhancing neurological function.

SECONDARY OUTCOMES:
Assessment of Intubation Requirement Using GCS and APACHE | participants were assessed within 24 hours from admission to the hospital
  This study investigates the requirement for intubation and mechanical ventilation among participants with acute carbamazepine poisoning using multiple clinical assessment tools, including the Glasgow Coma Scale (GCS) and Acute Physiology and Chronic Health Evaluation (APACHE). The GCS evaluates the level of consciousness based on eye opening, verbal response, and motor response, with lower scores indicating a higher likelihood of intubation and mechanical ventilation. The APACHE score assesses the severity of illness and predicts the need for respiratory support, with higher scores indicating an increased risk of respiratory failure and the requirement for intervention.
Length of Intensive Care Unit (ICU) Stay | Participants will be monitored throughout their hospitalisation period, and the length of their ICU stay will be recorded from date of randomization until the date of last documented progression up to one month
  This study evaluates the length of stay in the Intensive Care Unit (ICU) among participants with acute carbamazepine poisoning. The length of the ICU stay is defined as the duration from the time of admission to the ICU to discharge from the ICU in days. Participants will be monitored throughout their hospitalisation period, and the length of their ICU stay will be recorded. The study aims to assess the impact of SMOF lipid administration on the duration of ICU stays, providing insights into its effectiveness in optimising resource utilisation and patient management. Understanding the factors influencing the length of the ICU stay may contribute to improved healthcare delivery and patient outcomes in acute carbamazepine poisoning.
length of hospital stay | Participants will be monitored throughout their hospitalisation period, and the length of their hospital stay will be recorded from date of randomization until the date of last documented progression up to one month
  This study evaluates the length of stay in the hospital among participants with acute carbamazepine poisoning. The length of stay is defined as the duration from the time of admission to the hospital to discharge from the hospital in days. Participants will be monitored throughout their hospitalisation period, and the length of their hospital stay will be recorded. The study aims to assess the impact of SMOF lipid administration on the duration of hospital stays, providing insights into its effectiveness in optimising resource utilisation and patient management. Understanding the factors influencing length of stay may contribute to improved healthcare delivery and patient outcomes in acute carbamazepine poisoning.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Sheta, professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

REFERENCES:
- [Background] Zyoud SH, Waring WS, Al-Jabi SW, Sweileh WM, Rahhal B, Awang R. Intravenous Lipid Emulsion as an Antidote for the Treatment of Acute Poisoning: A Bibliometric Analysis of Human and Animal Studies. Basic Clin Pharmacol Toxicol. 2016 Nov;119(5):512-519. doi: 10.1111/bcpt.12609. Epub 2016 May 20. PMID 27098056
- [Background] Karaman K, Turkdogan KA, Deniz AT, Canakci SE. Which is the best in carbamazepine overdose? Clin Case Rep. 2017 Aug 22;5(10):1612-1615. doi: 10.1002/ccr3.1118. eCollection 2017 Oct. PMID 29026556
- [Background] Jaffal K, Chevillard L, Megarbane B. Lipid Emulsion to Treat Acute Poisonings: Mechanisms of Action, Indications, and Controversies. Pharmaceutics. 2023 May 3;15(5):1396. doi: 10.3390/pharmaceutics15051396. PMID 37242638
- [Background] Taftachi F, Sanaei-Zadeh H, Sepehrian B, Zamani N. Lipid emulsion improves Glasgow coma scale and decreases blood glucose level in the setting of acute non-local anesthetic drug poisoning--a randomized controlled trial. Eur Rev Med Pharmacol Sci. 2012 Mar;16 Suppl 1:38-42. PMID 22582483